CLINICAL TRIAL: NCT03063307
Title: Effectiveness of Silver Diamine Fluoride in Arresting Dental Caries in Deciduous Molars: a Controlled and Randomized Clinical Trial
Brief Title: Effectiveness of Silver Diamine Fluoride in Arresting Dental Caries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Ana Lúcia Vollú, Postgraduate student,, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: silverdiamine
Record Dates: First submitted 2017-02-15; First posted 2017-02-24 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Dental Caries in Children
Keywords: Tooth, Deciduous; Dental Caries; Glass Ionomer Cements; Dental Atraumatic Restorative Treatment; Cariostatic Agents; Fluorides
MeSH Terms: conditions — Dental Caries | interventions — Dental Atraumatic Restorative Treatment; Glass Ionomer Cements; Ketac Molar Easymix; silver diamine fluoride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atraumatic Restorative Treatment (Active Comparator)
  Interventions: Procedure: Atraumatic Restorative Treatment
- Silver Diamine Fluoride (Experimental)
  Interventions: Other: Silver Diamine Fluoride

INTERVENTIONS:
Procedure: Atraumatic Restorative Treatment
  Other Names: ART; Glass Ionomer Cements; Ketac Molar Easymix
  Arms: Atraumatic Restorative Treatment
Other: Silver Diamine Fluoride
  Other Names: SDF; SDF 30%; Cariostop 30% Biodinâmica
  Arms: Silver Diamine Fluoride

SUMMARY:
The present study aims to evaluate, through a controlled clinical randomized study,the effectiveness of silver diamine fluoride in arresting dentin caries lesions in primary molars when compared to atraumatic restorative treatment.

DETAILED DESCRIPTION:
The present controlled clinical randomized study aiming at evaluating the effectiveness of silver diamine fluoride (SDF) in arresting dentin caries lesions on the occlusal surface of primary molars when compared to atraumatic restorative treatment (ART). For this, 118 healthy children aged 2-5 years with at least one active dentin carious lesion, with no signs of pain or pulp involvement. The participants will be allocated randomly to one of two treatment groups: (1) Test Group - SDF and (2) Control Group - ART. The International Caries Detection and Assessment System (ICDAS) will be used to determine caries diagnosis and activity. In both groups, the guardians and children will receive oral hygiene instructions and will be advised about eating habits and fluoride dentifrice use.The clinical success will be verified through examinations performed by a blinded operator, after 3, 6 and 12 months, with clinical evaluations to detect caries arresting, representing the primary outcome of the study.

ELIGIBILITY:
Inclusion Criteria:

* CHILDREN

  * aged 2 to 5 years;
  * who are in good general health;
  * have at least one active dentin carious lesion on the occlusal surface of primary molars corresponding to ICDAS codes 5 or 6.

Exclusion Criteria:

* CHILDREN

  * with systemic or neurological diseases;
  * whose families intend to move from Rio de Janeiro next year;
  * with a history of allergy to silver or any substance present in the different materials to be used for treatment.

TEETH

* with spontaneous or provoked pain, dental mobility or radiographic signs of involvement or possible pulp involvement;
* shows possible pulp involvement by radiographic examination

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Caries arresting | The follow-up oral examinations will be conducted every 3 months for 48 months totally
  The main outcome of the study will be the observation of the proportion of arrested caries lesions in the test group, compared to the control group.

SECONDARY OUTCOMES:
Duration of the intervention visit | 1 year
  Time (in minutes) spent on each type of intervention (DFP x ART)
Cost | 1 year
  The cost of each treatment will be recorded and compared to each other
Aesthetic perception and treatment satisfaction | First appointment, 3,6 and 12 months after treatment.
  Information on aesthetic perception will be obtained through a questionnaire, addressed to parents / guardians.
Anxiety | From allocation up to two weeks.
  A facial imaging scale will be used to assess the degree of anxiety of children 3 years of age or older. before and after first exam and treatment appointments.
Quality of life assessment | First appointment,15 days and 3 months after treatment.
  Information about quality of life will be obtained through the questionnaire Brazilian Early Childhood Oral Health Impact Scale (B-ECOHIS), addressed to parents / guardians.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Lucia Vollu, MSD Student, Principal Investigator — Universidade Federal Fluminense
Locations (1):
- Departamento de Odontopediatria e Ortodontia da UFRJ, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodrigues GF, Vollu AL, Vargas TR, Kamp LMK, da Cunha Costa T, Cruz LR, Luiz RR, Barja-Fidalgo F, Fonseca-Goncalves A. Efficacy of 30% silver diamine fluoride compared to atraumatic restorative treatment in arresting dentin caries lesions in preschoolers: a randomized clinical trial. Clin Oral Investig. 2024 Dec 6;29(1):3. doi: 10.1007/s00784-024-06081-8. PMID 39641816